CLINICAL TRIAL: NCT04329221
Title: Calcipotriol Plus 5-Flourouracil Immunotherapy Before Transplantation for Skin Cancer Prevention in Organ Transplant Recipients
Brief Title: Immunotherapy Before Transplantation for Skin Cancer Prevention in Organ Transplant Recipients
Status: Withdrawn | Phase: Phase 2 | Type: Interventional
Why Stopped: The study was withdrawn due to lack of financial support.
Sponsor: Massachusetts General Hospital (Other)
Collaborators: Washington University School of Medicine (Other)
Responsible Party: Principal Investigator, Shadmehr Demehri, MD, PHD, Massachusetts General Hospital
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Prevention
Other Study IDs: 2019P003401
Record Dates: First submitted 2020-03-30; First posted 2020-04-01 (Actual); Last update posted 2025-05-07 (Actual); Status verified 2025-05

CONDITIONS: Cutaneous Squamous Cell Carcinoma; Actinic Keratoses; Skin Cancer; Organ Transplant Recipients; Immunotherapy
Keywords: Calcipotriol ointment; 5-FU cream; Squamous Cell Carcinoma; Actinic Keratoses; Organ Transplant Recipients; Prevention; Immunotherapy
MeSH Terms: conditions — Keratosis, Actinic; Skin Neoplasms; Carcinoma, Squamous Cell | interventions — Petrolatum; Fluorouracil

STUDY DESIGN:
Intervention Model Description: Parallel assignment
Who Masked: Participant, Care Provider, Investigator
Masking Description: All participants, care giver and investigators measuring or analyzing the experimental data will be blinded to the interventions. Tissue samples collected will be labeled with 3-digit unique IDs and de-identified before studying in PI's lab. The study investigator will collect AK/skin samples and label them based on the study ID (e.g. "201") without compromising their blinded status. All the study records/photographs will be kept in a locked office or password-protected computer that is only accessible by the members of the research team.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (2):
- Topical Calcipotriol ointment plus 5-Fluorouracil cream (Experimental): Topical Calcipotriol 0.0025% ointment plus 5-Fluorouracil 2.5% cream will be administered by the participants to their face, scalp and upper extremities twice a day for 6 consecutive days.
  Interventions: Drug: Calcipotriol Only Product in Cutaneous Dose Form; Drug: Topical 5FU
- Topical vaseline plus 5-Fluorouracil 2.5% cream (Placebo Comparator): Topical Vaseline plus 5-Fluorouracil 2.5% cream will be administered by the participants to their face, scalp and upper extremities twice a day for 6 consecutive days.
  Interventions: Drug: Vaseline; Drug: Topical 5FU

INTERVENTIONS:
Drug: Calcipotriol Only Product in Cutaneous Dose Form — Calcipotriol (Calcipotriene) is a form of vitamin D. It works by inducing thymic stromal lymphopoietin cytokine expression in the skin.
  Other Names: Topical Calcipotriol ointment
  Arms: Topical Calcipotriol ointment plus 5-Fluorouracil cream
Drug: Vaseline — Placebo
  Other Names: Petrolatum
  Arms: Topical vaseline plus 5-Fluorouracil 2.5% cream
Drug: Topical 5FU — 5-FU is a chemotherapy that causes the death of proliferating tumor cells. Topical preparation of this drug is being used.
  Other Names: Topical 5-fluorouracil

SUMMARY:
This clinical trial aims to investigate the efficacy of Calcipotriol ointment combined with 5-fluorouracil cream as an immunotherapy for actinic keratosis in Organ Transplant Recipients (OTRs) before transplantation and determine whether it can prevent cutaneous squamous cell carcinoma (SCC) in OTRs post-transplant.

DETAILED DESCRIPTION:
The main goal of this investigator-initiated clinical trial is to determine the efficacy of topical calcipotriol combined with 5-flourouracil (5-FU) treatment in organ transplant candidates with precancerous skin lesions called actinic keratoses (AKs) with a history of skin cancer in order to prevent squamous cell carcinoma (SCC) development after transplantation. SCC is the most common cutaneous malignancy seen after transplantation, with a 65-250 fold greater incidence in organ transplant recipients (OTRs) compared to the general population. This increased risk is due to the systemic immunosuppression caused by anti-rejection medications, which are indispensable for protecting against allograft loss. Previously, we have demonstrated the high efficacy of topical calcipotriol plus 5-FU immunotherapy for AKs on the face and scalp in significantly reducing the risk of SCC development within 3 years post-treatment in immunocompetent patients. This SCC risk reduction is accompanied by the induction of robust T cell immunity and TRM cell formation against AKs. Calcipotriol is a low calcemic vitamin D analogue that is FDA-approved for the treatment of psoriasis. Topical 5-FU is a chemotherapy that is the standard treatment for AKs. Our previous research demonstrates the synergistic impact of calcipotriol in combination with 5-FU on a robust T cell immunity against early skin carcinogenesis in immunocompetent patients. Therefore, we aim to determine the efficacy of this immunotherapy before transplantation in reducing the risk of SCC post-transplant despite the immunosuppressive medications.

ELIGIBILITY:
Inclusion Criteria:

* Solid organ transplant candidates with AKs and a history of non-melanoma skin cancer. The target population includes the patients who are undergoing kidney, lung, liver and heart transplantations.
* Presence of four to fifteen clinically typical, visible, and discrete AKs in 25 cm2 on any of the four anatomical sites: scalp, face, right upper extremity and left upper extremity.
* The period between the first visit and transplantation is minimum 4 weeks and maximum 12 months.
* Age of at least 18 years
* Ability and willingness of the patient to participate in the study (Informed consent will be obtained)

Exclusion Criteria:

* Treatment area is within 5 cm of an incompletely healed wound or a suspected basal cell or squamous cell carcinoma.
* Treatment area contained hypertrophic and hyperkeratotic lesions, cutaneous horns, or lesions that had not responded to repeated cryotherapy.
* Patients with history of hypercalcemia or vitamin D toxicity.
* Female participants must be either of non-reproductive potential (i.e., post-menopausal by history of age > 50 years old and no menses for >1 year without an alternative medical cause; OR history of hysterectomy, history of bilateral tubal ligation, or history of bilateral oophorectomy) OR must have a negative serum pregnancy test within 7 days prior to study registration.
* Patients with DPD (Dihydropyrimidine Dehydrogenase) deficiency (due to their higher risk of 5-FU toxicity).

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2029-01 (Estimated); Study Completion 2030-01 (Estimated)

PRIMARY OUTCOMES:
The changes in the percentage of participants with new SCC on treated anatomical sites in OTRs | Year 2 post-transplant
  The changes in the percentage of participants with new SCC on treated anatomical sites quantified based on participants' medical records, photographs and pathology results after transplantation in test versus control group.

SECONDARY OUTCOMES:
The percent change in baseline number of AKs on the treated anatomical sites in OTRs. | 8 weeks after treatment
  The percent change in baseline number of AKs on the treated anatomical sites in post-transplant OTRs quantified based on participants' medical records and photographs after transplantation in test versus control group
The changes in TSLP, CD3+, CD4+ and CD8+ TRM cell infiltrates and other immune factors/cells in the AK and normal skin | at one day after 6-day treatment and at one year post-transplant.
  The changes in TSLP, CD3+, CD4+ and CD8+ TRM cell infiltrates and other immune factors/cells in the AK and normal skin in test versus control group after treatment and transplantation compared to before treatment.
The changes in immune infiltrate in any SCC that develops after treatment | for up to 4 years post-transplant
  The changes in immune infiltrate in any SCC that develops after calcipotriol plus 5-FU versus Vaseline plus 5-FU treatment
The changes in SCC prevention (SCC number) on the untreated anatomical sites (i.e., trunk and lower extremities) of OTRs | at one, two and four years post-transplant.
  The changes in efficacy of a twice daily 6-day treatment with topical calcipotriol plus 5-FU (test) versus Vaseline plus 5-FU (control) before transplantation in preventing SCC on the untreated anatomical sites (i.e., trunk and lower extremities) of OTRs.
The changes in erythema extent and intensity scores of the treated anatomical sites | at one day after the completion of a 6-day treatment.
  The changes in erythema extent and intensity scores of the treated anatomical sites after treatment in test versus control group. Treated skin will be evaluated for any sign of irritation including erythema, crusting or ulceration using a clinical erythema scale.
Number of Participants with Treatment Related Adverse Events | From the start of treatment until 30 days after the end of treatment, up to 2 months
  Adverse events will be assessed including any local skin reactions like itching and rash.
Number of participants with any proven rejection of the graft in OTRs | From the start of treatment until 30 days after the end of treatment
  Number of participants with any biopsy proven acute rejection of the graft after treatment with calcipotriol plus 5-FU compared to test group
The changes in response to treatment (AK and SCC number) between treated anatomical sites | at one day after treatment and one year after transplantation.
  The changes in response to topical calcipotriol plus 5-FU versus Vaseline plus 5-FU between treated anatomical sites

CONTACTS AND LOCATIONS:
Overall Officials: Shadmehr Demehri, MD/PHD, Principal Investigator — Massachusetts General Hospital
Locations (2):
- United States (2):
  - Massachusetts General Hospital, Boston, Massachusetts
  - Barnes-Jewish Hospital, St Louis, Missouri

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Cunningham TJ, Tabacchi M, Eliane JP, Tuchayi SM, Manivasagam S, Mirzaalian H, Turkoz A, Kopan R, Schaffer A, Saavedra AP, Wallendorf M, Cornelius LA, Demehri S. Randomized trial of calcipotriol combined with 5-fluorouracil for skin cancer precursor immunotherapy. J Clin Invest. 2017 Jan 3;127(1):106-116. doi: 10.1172/JCI89820. Epub 2016 Nov 21. PMID 27869649
- [Background] Rosenberg AR, Tabacchi M, Ngo KH, Wallendorf M, Rosman IS, Cornelius LA, Demehri S. Skin cancer precursor immunotherapy for squamous cell carcinoma prevention. JCI Insight. 2019 Mar 21;4(6):e125476. doi: 10.1172/jci.insight.125476. eCollection 2019 Mar 21. PMID 30895944